CLINICAL TRIAL: NCT02576392
Title: Reducing the Use of Opioid Therapy Following Orthopedic Surgery: A Randomized Controlled Trial
Brief Title: FDA: Lowering Orthopedic Opioid Dosing (FLOOD)
Acronym: FLOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FDA BAA HHSF223201400146C
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Informational letter mailed approximately 2 weeks prior to surgery, informational letter mailed approximately 2 weeks post surgery, pharmacist call if refill opioid medicine more than 28 days after surgery
  Interventions: Behavioral: Intervention
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Intervention — Intervention consisted of a mailing 2 weeks prior to surgery, another 2 weeks post surgery, and a pharmacist intervention if a refill of opioid medication was requested within 90 days of surgery.
  Arms: Intervention

SUMMARY:
This randomized trial evaluates an intervention to minimize use of opioids following total hip and total knee replacement. Half the participants will receive an intervention (mailed educational materials, followed by a pharmacist call), and half will receive usual care.

DETAILED DESCRIPTION:
Surgeons and anesthesiologists prescribe opioids and other analgesic medications for acute, post-surgical pain. Recent studies have reported that some patients persist in taking opioids for months beyond the surgery. While opioids are commonly used for pain management following surgery, patients and their providers often don't have a planned method to optimize opioid exposure. This can lead to patients entering a cycle of opioid use that is difficult to manage, because, as opioid exposure is continued, pain relief is reduced and side effects increase. The investigators' study is aimed at reducing opioid exposure following total hip and total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* total hip replacement or total knee replacement
* 1 year membership with KPNW prior to enrollment

Exclusion Criteria:

* managed by pain clinic, in other pain management trial
* patients at low risk of persistent opioid use

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2015-07-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Average morphine equivalents | 90 days
  post surgery use of opioids

CONTACTS AND LOCATIONS:
Overall Officials: David H Smith, RPh, PhD, Principal Investigator — Kaiser Permanente NW

IPD SHARING:
Plan to Share IPD: No